CLINICAL TRIAL: NCT07214233
Title: Youth Empowerment and Safety Intervention for Systems-involved Sexual and Gender Minority Youth at Risk of Suicide
Brief Title: Youth Empowerment and Safety Intervention
Acronym: YES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: FrontLine Service (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY20241289; 1R34MH134912-01A1 (NIH)
Record Dates: First submitted 2025-10-07; First posted 2025-10-09 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Suicide; Self-Injurious Behavior
Keywords: Self-injurious thoughts and behaviors (SITB); Peer Support Specialist (PSS); Behavioral health; adolescent; LGBTQ; Juvenile Justice; Foster Care; Crisis Response
MeSH Terms: conditions — Suicide; Self-Injurious Behavior; Behavior | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-implementation Period (Active Comparator): Behavioral health treatment as usual
  Interventions: Behavioral: Treatment as Usual
- Post-implementation Period (Experimental): Behavioral health treatment as usual + referral to and connection with Peer Support Services
  Interventions: Behavioral: Peer Support Services (PSS)

INTERVENTIONS:
Behavioral: Treatment as Usual — Behavioral health services (treatment as usual)
  Arms: Pre-implementation Period
Behavioral: Peer Support Services (PSS) — Behavioral health services (treatment as usual) along with referral to and utilization of Peer Support Specialist services
  Arms: Post-implementation Period

SUMMARY:
This clinical trial will implement and evaluate the feasibility, acceptability, and initial impact of Peer Support Specialist (PSS) services for public system-involved sexual and gender minority (lesbian, gay, bisexual, queer and/or transgender) youth (SGMY) at risk of suicide.

DETAILED DESCRIPTION:
A sharp increase in U.S. youth mental health problems coupled with the national shortage in child behavioral health clinicians has identified peer providers as a cost- and impact-effective solution. Peer Support Specialists (PSS), paraprofessionals with lived experience who provide mutual and structured support, have been found to be effective in improving client engagement in mental health services. The study proposes to evaluate the feasibility, acceptability, and initial impact of a multi-level intervention, Youth Empowerment & Safety (YES), comprised of two coordinated components: 1) system-level improved identification and referral (I/R) of self-injurious thoughts and behaviors (SITB) among sexual and gender minority youth (SGMY), and 2) introduction of an SGMY-tailored support PSS to enhance engagement and support with behavioral health treatment and other support services.

ELIGIBILITY:
Child Inclusion Criteria:

* 12-17 years of age
* Self-identify as a sexual or gender minority (SGM)
* Involved in one or more system: juvenile justice, child welfare, and/or community-based mental health
* Personal experience with self-injurious thoughts and behaviors (SITB)
* English speaking
* Willing and able to provide informed assent

Child Exclusion Criteria:

* Less than 12 or greater than 17 years of age (0-11 or 18 and over)
* Do not self-identify as a sexual or gender minority (SGM)
* Not involved in the juvenile justice, child welfare, and/or community-based mental health systems
* No personal experience with self-injurious thoughts and behaviors (SITB)
* Not English speaking
* Unwilling and/or unable to provide informed assent

Caregiver Inclusion Criteria:

* 18-80 years of age
* Primary Caregiver of youth who meet child inclusion criteria listed above
* English speaking
* Willing and able to provide informed consent

Caregiver Exclusion Criteria:

* Less than 18 or greater than 80 years of age (0-17 or 81 and over)
* Not the Primary Caregiver of youth who meet child inclusion criteria listed above
* Not English speaking
* Unwilling and/or unable to provide informed consent

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Youth-level changes in Recovery | Baseline, Post-Intervention 3 Month, and Post Intervention 6 Month
  The researchers will compare the change in treatment engagement as quantified by total score on two separate subscales of the Questionnaire about the Process of Recovery (the QPR). The QPR is a 22-item measure developed from service users' accounts of recovery in collaboration with local service users. Each item is scored using a 5-point Likert scale ranging from 0 (disagree strongly) to 4 (agree strongly). There are two subscales: 1) intrapersonal tasks involved in recovery (17 items, range 0-68) and 2) interpersonal factors that facilitate recovery (5 items, range 0-20) with higher scores indicating increased recovery on both subscales.
Youth Level Changes in Self-injurious thoughts and behaviors | From enrollment (baseline), to 3- and 6 months follow ups post treatment at the end of 8-12 weeks.
  The researchers will compare changes in suicidal ideation, planning, attempt and non-suicidal self-harm in a group of pre-intervention (nonrandomized) youth to post-intervention (nonrandomized youth) using the Columbia Suicide Severity Rating Scale (C-SSRS), a widely used and well-validated measure of suicidal ideation, planning, attempt, and non-suicidal self-harm.

SECONDARY OUTCOMES:
Patient Health Questionnaire - Depression Scale - PHQ-9 | Study enrollment (baseline) and 3- and 6-month follow-ups
  The Patient Health Questionnaire - Depression Scale (PHQ-9) is a validated measure of depression consisting of nine questions that assess the severity of depressive symptoms over the past two weeks. Each item is scored using a 4-point Likert scale ranging from 0 (Not at all) to 3 (Nearly every day). The scale provides a cumulative score (range from 0-27) with higher scores suggesting more severe depressive symptoms.
Youth level changes in minority stress | baseline, 3- month post, 6-month follow up
  The researchers will assess changes in minority stress, as measured by the Adolescent Minority Stress Inventory. This is a 26-item measure of minority stressors experienced by LGBTQ+ youth in the past 30 days utilizing a binary Yes/No scale (yes = 1, no = 0). The scale provides a cumulative score (range from 0-30) with higher scores suggesting higher stress.
Youth Level Changes in Perceived Parent Acceptance | baseline, 3-month post, 6 month follow up
  The Family Acceptance Measure is a 6-item measure of youths' perception of accepting and rejecting attitudes and behaviors of LGBTQ+ youth. Each item is scored using a 4-point Likert scale ranging from 0 (Never) to 3 (Often). The scale provides a cumulative score (range from 0-18) with higher scores suggesting less familial acceptance.

CONTACTS AND LOCATIONS:
Overall Officials: Dana M. Prince, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
This is a community participatory research design. Members of the Learning Collaborative will be involved in the final decision about IPD sharing.

REFERENCES:
- [Background] Prince DM, Ray-Novak M, Gillani B, Peterson E. Sexual and Gender Minority Youth in Foster Care: An Evidence-Based Theoretical Conceptual Model of Disproportionality and Psychological Comorbidities. Trauma Violence Abuse. 2022 Dec;23(5):1643-1657. doi: 10.1177/15248380211013129. Epub 2021 May 4. PMID 33942681
- [Background] Gillani B, Prince DM, Ray-Novak M, Feerasta G, Jones D, Mintz LJ, Moore SE. Mapping the Dynamic Complexity of Sexual and Gender Minority Healthcare Disparities: A Systems Thinking Approach. Healthcare (Basel). 2024 Feb 6;12(4):424. doi: 10.3390/healthcare12040424. PMID 38391800
- [Background] Prince, D. M., Ray-Novak, M*. Tossone, K., Peterson, E.*, Gillani, B.*, & Mintz, L. (2024). Psychological comorbidities and suicidality in sexual and gender minority foster youth. Children and Youth Services Review, 156 (2024): 107379.
- [Background] Prince DM, Schuler MS, Lewis K, Munson MR, Blashill AJ, Hovmand PS. Opportunities to Address Health Disparities in Suicidality for Sexual and Gender Minority Youth in Public Systems. Mental Health Sci. 2025 Mar;3(1):10.1002/mhs2.100. doi: 10.1002/mhs2.100. Epub 2024 Dec 19. No abstract available. PMID 41367936